CLINICAL TRIAL: NCT06698354
Title: Cost-Effectiveness Analysis of a Virtual Reality-Assisted Hypnotherapy Program on Quality of Life in Patients with Chronic Low Back Pain: a Multicenter, Randomized, Prospective, Comparative, Open-Label, Parallel-Group Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, TUĞBA ŞAHBAZ, Associate Professor, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-66291034-202.3.02-6546
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain; Low Back Pain; Chronic Low Back Pain (CLBP)
Keywords: hypnotherapy; virtual reality
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality-Assisted Hypnotherapy+Physiotherapy Group (Experimental): Participants in this arm will undergo a conventional physical therapy program for 3 weeks (15 sessions) supervised by physiotherapists. Additionally, during each physical therapy session, participants will receive a 20-minute Virtual Reality (VR)-assisted hypnotherapy session using the HypnoVR software.
  Interventions: Device: Virtual Reality-Assisted Hypnotherapy
- Standard Treatment Group (Active Comparator): Participants in this arm will undergo a conventional physical therapy program for 3 weeks (15 sessions) supervised by physiotherapists.
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Device: Virtual Reality-Assisted Hypnotherapy — Virtual Reality-Assisted Hypnotherapy utilizes HypnoVR software delivered through VR glasses to provide a relaxing virtual environment. The intervention is integrated into a standard physical therapy program, with participants receiving 20-minute VR-assisted hypnotherapy sessions during each of the 15 supervised physical therapy sessions over a 3-week period. This approach aims to improve pain management, quality of life, and adherence to treatment in patients with chronic low back pain.
  Arms: Virtual Reality-Assisted Hypnotherapy+Physiotherapy Group
Other: Standard Physical Therapy — Participants in the control group will undergo a standard physical therapy program focused on the cervical region, consisting of 15 sessions over 3 weeks. Each session will be supervised by physiotherapists in a clinical setting and will include traditional physical therapy techniques such as therapeutic exercises
  Arms: Standard Treatment Group

SUMMARY:
This randomized, prospective study aims to evaluate the effectiveness and cost-efficiency of a Virtual Reality (VR)-assisted hypnotherapy program on quality of life in patients with chronic low back pain. The study compares a VR-assisted hypnotherapy group to a standard treatment group. Both groups will undergo a conventional physical therapy program supervised by physiotherapists for 3 weeks (15 sessions). The VR-assisted hypnotherapy group will receive additional sessions utilizing the HypnoVR software, which delivers relaxing virtual environments. Outcomes will be assessed immediately after treatment, at 1 month, and at 3 months post-treatment. Primary endpoints include pain reduction measured by the Visual Analog Scale (VAS). Secondary endpoints include functionality, quality of life, anxiety, depression, sleep quality, healthcare costs, and treatment adherence. Statistical analyses will determine the efficacy and economic impact of this innovative therapy for chronic low back pain management.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 80 years.
* Chronic neck pain lasting for more than 3 month

Exclusion Criteria:

* Presence of newly developed neurological deficits.
* Existence of comorbid neurological diseases.
* Medical history unsuitable for the use of virtual reality (VR) glasses (e.g., visual impairment, epilepsy).
* Pregnancy.
* Changes in medication for chronic pain management within the last three months (e.g., Pregabalin, Gabapentin, Duloxetine, etc.).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Assessed at baseline, immediately after treatment (3 weeks), and at 1- and 3-month follow-ups.
  The primary outcome is the percentage change in pain intensity, measured using the Visual Analog Scale (VAS). A reduction of ≥30% in the VAS score from baseline is considered clinically significant.

SECONDARY OUTCOMES:
Change in Functional Status | Baseline, post-treatment (3 weeks), and at 1- and 3-month follow-ups.
  Functional status will be assessed using the Roland-Morris Disability Index.
Change in Quality of Life | Baseline, post-treatment (3 weeks), and at 1- and 3-month follow-ups.
  Quality of life will be measured using the EQ-5D-5L questionnaire.
Reduction in Analgesic Use | Baseline and weekly throughout the 3-month follow-up period.
  The number of days per week participants use nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen for pain management will be recorded.
Change in Anxiety and Depression Levels | Baseline, post-treatment (3 weeks), and at 1- and 3-month follow-ups.
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS).
Reduction in Healthcare Utilization | Assessed retrospectively at baseline and at the 3-month follow-up.
  Healthcare utilization, including the number of clinic visits (Family Medicine, Physical Therapy, Orthopedics) and cervical imaging (X-ray, MRI), will be recorded for the 3 months prior to and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Beykent University Faculty of Medicine, Physical Therapy Unit, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Menekseoglu AK, Asik HK, Sahbaz T, Is EE. Mind over pain: VR-based hypnotherapy for chronic non-specific low back pain - a randomised controlled trial. Ir J Med Sci. 2025 Nov 10. doi: 10.1007/s11845-025-04158-1. Online ahead of print. PMID 41212507
- See also: Related Info — https://hypnovr.io/en/